CLINICAL TRIAL: NCT03600272
Title: Comparison of Combined Spinal-epidural Analgesia Versus Epidural Analgesia During Labor
Brief Title: Comparison of Combined Spinal-epidural Analgesia Versus Epidural Analgesia for Pain Management During Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Deng Dongrui (Other)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor-Investigator, Deng Dongrui, Professor, Chief doctor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ-C20180711
Record Dates: First submitted 2018-07-10; First posted 2018-07-26 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Labor Long; Labor Pain; Labor Fetal Anoxia
Keywords: Combined spinal-epidural analgesia; Epidural analgesia; Labor duration
MeSH Terms: conditions — Labor Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: Participants who request neuraxial labor analgesia are randomly assigned into two groups by a computer-generated random number table using Excel. One group received combined spinal-epidural analgesia during labor, the other group received epidural analgesia during labor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One anesthetist who were not involved with clinical care or data collection performed the randomization procedure and the neuraxial block according to the group allocation. The other anesthetist blinds to the procedure preform the analgesia management after neuraxial block. This anesthetist and the obstetrician, the midwives, the patients , the outcomes collector and assessor are all blind to group allocation throughout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined spinal-epidural analgesia (Experimental): The combined spinal epidural analgesia technique was used to maintain analgesia for parturients in the combined spinal-epidural analgesia group. First, the investigator injected a dose of 5 ug sufentanil into cerebrospinal fluid. If no adverse effects were observed 10 minutes after the first dose, the parturient then received mixed liquids of 0.075% ropivacaine and 0.2ug/ml sufentanil citrate through a patient-controlled epidural analgesia (PCA) pump, which provided patients themixed solution at 8-10ml/h to optimize their pain relief until the delivery of neonates.
  Interventions: Procedure: Combined spinal-epidural analgesia
- Epidural analgesia (Other): The epidural analgesia technique was used to maintain analgesia for parturients in the epidural analgesia group, which involved placing a thin catheter through a needle inserted into the epidural space. First, the investigator injected a test dose of 5ml 1% lidocaine through it. If not adverse effects were observed 10 minutes after the test dose, the parturient then received a bolus injection of an initial dose of 8-10 ml mixed liquids of 0.075% ropivacaine and 0.2ug/ml sufentanil citrate. We then connected the catheter with a patient-controlled epidural analgesia (PCA) pump, which provided patients the same mixed solution at 8-10ml/h to optimize their pain relief until the delivery of neonates.
  Interventions: Procedure: Epidural analgesia

INTERVENTIONS:
Procedure: Combined spinal-epidural analgesia — Combined spinal-epidural analgesia during labor is a labor analgesia technique which reported maybe associate with a shorter labor duration compared to the traditional epidural labor analgesia.
  Arms: Combined spinal-epidural analgesia
Procedure: Epidural analgesia — Epidural analgesia is a well-accepted technique using for pain relief during labor.
  Arms: Epidural analgesia

SUMMARY:
The investigators want to compare the safety and efficacy between the combined spinal-epidural analgesia and epidural analgesia during labor.

DETAILED DESCRIPTION:
Participants who request neuraxial labor analgesia are randomized to receive combined spinal-epidural analgesia or epidural analgesia during labor. The investigators collect the data on the duration of three stages of labor, the mode of delivery, neonatal Apgar scores, VAS scores, modified Bromage scores.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women at term (37 to 42 weeks of gestation), vertex presentation, singleton pregnancy who desired vaginal delivery were eligible to participate.

Exclusion Criteria:

* Contraindications to neuraxial techniques such as clinically significant coagulopathy and increased intracranial pressure, and patients with preterm labor, multiple pregnancies, non-vertex presentation, cephalopelvic disproportion and severe obstetric complications

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-20 (Estimated); Primary Completion 2018-11-20 (Estimated); Study Completion 2019-07-20 (Estimated)

PRIMARY OUTCOMES:
Labor duration | At the end of delivery
  Duration of three stages of labor

SECONDARY OUTCOMES:
The mode of delivery | At the end of delivery
  Including spontaneous vaginal delivery, vacuum- and forceps-assisted delivery, cesarean delivery
1 minute and 5 minutes Apgar scores | 1 min after delivery, 5 min after delivery.
  Neonatal Apgar scores at the first and fifth minute.The score indicates the infant s' conditions, including heart rate, breathing, muscle tone, reflex response, color. Each characteristic is given an individual score; two points for each of the five categories if all is completely well; then all scores are totaled. The score is from 0 to 10.
Visual Analogue Scores(VAS) | At 5min before analgesia; at 5min, 15min, 30min, 1h after the first dose of analgesic drugs； at cervical dilation of 3cm , 6cm and 10cm; at the time of birth of infant; at the time of delivery of placenta.
  VAS is the most common pain scale for quantification. The score is higher, the patient will be more painful. That will indicate if the analgesia is effective. Visual analog scale (VAS) ranging from 0 to 10 (with 10 representing the worst pain imaginable) to measure the degree of pain for participants.
Modified Bromage scores | At 5min before analgesia; at 5min, 15min, 30min, 1h after the first dose of analgesic drugs； at the cervical dilation of 3cm , 6cm and 10cm; at the time of birth of infant; at the time of delivery of placenta.
  The modified Bromage score is the most frequently used measure of motor block. In this scale, the intensity of motor block is assessed by the patient's ability to move their lower extremities(0: no motor paralysis; 1: inability to raise extended leg, but able to move knee and foot; 2: inability to raise extended leg and to move knee, but able to move foot; 3: inability to raise extended leg or to move knee and foot).

CONTACTS AND LOCATIONS:
Overall Officials: Haiyi Liu, M.D., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided